CLINICAL TRIAL: NCT05181280
Title: Moms on Media Study: Testing the Influence of Social Media on the Health Behaviours of Mothers During the Postpartum Period
Brief Title: Moms on Media Study
Acronym: MOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Canadian Foundation for Dietetic Research (CFDR) (Other)
Responsible Party: Principal Investigator, Lisa Tang, Principal Investigator, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 054798
Record Dates: First submitted 2021-12-08; First posted 2022-01-06 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants are randomized into either the intervention group (body image messaging) or control group (infant feeding messaging).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Treatment: Standardized body image messaging targeting mothers. Following a similar model that has been used in previous studies testing the effect of traditional media exposure on body image and disordered eating behaviour, participants randomized to the treatment condition will have 1 exposure session per day over 5 days. Each exposure session will consist of 15 social media body message posts. Body image messaging targeting mothers will consist of mothers with "ideal" postpartum bodies and captions trending over the past 24 months.
  Interventions: Other: Intervention Group
- Control (Placebo Comparator): Control: Standardized infant feeding tips messaging. Participants randomized to the control will have 1 exposure session/day over 5 days. Each exposure will consist of 15 social media posts on infant feeding tips.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention Group — Exposure session will consist of 15 social media "ideal body" message posts.
  Arms: Intervention
Other: Control Group — Exposure will consist of 15 social media posts on infant feeding tips.
  Arms: Control

SUMMARY:
This research will explore the impact of digital technology, specifically social media, on the health behaviours of mothers in the postpartum period by conducting an experimental study to test the effect of social media messaging on body dissatisfaction, eating attitudes and behaviours, and physical activity intentions and behaviours among postpartum mothers. The primary objective is to determine the extent to which body image messaging targeting mothers, compared with the control, result in feelings of body dissatisfaction and poorer eating attitudes and behaviours, and increased physical activity intention immediately following the 5-day exposure period. The secondary objective is to determine the sustained impact of the body image messaging compared to control at 1-month follow-up.

DETAILED DESCRIPTION:
The postpartum period is a critical time for both maternal and child health. Body dissatisfaction is higher during the postpartum period compared to other periods of life and is strongly associated with disordered eating behaviours. Body dissatisfaction among mothers not only effects the health of mothers but can also negatively influence the eating attitudes and behaviours of their children.

Although research has shown that media images have a strong adverse influence of women's body dissatisfaction, most of this research has focused on traditional forms of media, such as magazines. Limited research has explored how messages and images on social media platforms, such as Facebook and Instagram, influence women's body dissatisfaction and disordered eating risk, and no studies have explored this association among mothers. This is a concern as nearly 90% of mothers use social media regularly. Thus, little is known about how the current media environment influences body dissatisfaction and eating behaviour during the postpartum period.

The proposed research will address this knowledge gap by conducting an experimental study to test the effect of social media messaging on body dissatisfaction, eating attitudes and behaviours, and physical activity intentions and behaviours among postpartum mothers. The primary objective is to determine the extent to which body image messaging targeting mothers, compared with the control, result in feelings of body dissatisfaction and poorer eating attitudes and behaviours, and increased physical activity intention immediately following the 5-day exposure period. The secondary objective is to determine the sustained impact of the body image messaging compared to control at 1-month follow-up.

This study will provide a much-needed understanding of the effect of digital technology on postpartum mothers' body dissatisfaction, eating attitudes and behaviours, and physical activity intentions and behaviours. Results will inform healthcare interventions, equipping clinicians with research-based evidence to support postpartum mothers in maintaining positive body image and healthy eating and physical activity attitudes and behaviours.

ELIGIBILITY:
Inclusion Criteria:

* Can respond to surveys in English
* Has a child 0-6 months old
* Owns a smartphone

Exclusion Criteria:

* History of anxiety or depression
* Taking pharmacological treatments for anxiety or depression

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
Change in Body Dissatisfaction at 5 days and 1 month | 5 days and 1 month
  Body dissatisfaction will be measured using the body satisfaction subscale from the Multidimensional Eating Disorder Inventory, a 9-item subscale that measures satisfaction with physical appearance. This subscale includes questions such as "I think my stomach is too big". This subscale has been validated among a diverse population of women, with good internal consistency. Response options are "never", "rarely", "sometimes", "often", "usually", and "always", and are coded as 1-6 respectively. Higher scores indicate higher levels of body dissatisfaction.

SECONDARY OUTCOMES:
Change in Eating Attitude at 5 days and 1 month | 5 days and 1 month
  Disordered eating attitudes will be measured using the validated Eating Attitudes Test (EAT-26), a 26 items scale that measures attitudes toward food, body, and eating. Response options for all questions are "never", "rarely", "sometimes", "often", "usually", "always" with higher scores indicating higher levels of disordered eating attitudes.
Change in Eating Behaviour at 5 days and 1 month | 5 days and 1 month
  Disordered eating behaviours will be measured using the Dutch Eating Behaviour Questionnaire (DEBQ), a 24-item questionnaire with 3 subscales that measures restrained eating, emotional eating (4-item version), and external eating. This well-established questionnaire was found to have good internal consistency among each of the 3 subscales (Cronbach's Alpha 0.80 - 0.95), has been used to examine the eating behaviours of mothers,49 and postpartum mothers, and has been validated among diverse populations. The DEBQ includes questions such as "how often do you refuse food and drink offered because you are concerned about your weight?". Response options range from never to very often are assigned a score between 1 and 5. Scored are summed for each of the subscales, with higher scores indicating more restrained eating, more emotional eating, and more external eating.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

REFERENCES:
- [Derived] Tang L, Tiggemann M, Haines J. #Fitmom: an experimental investigation of the effect of social media on body dissatisfaction and eating and physical activity intentions, attitudes, and behaviours among postpartum mothers. BMC Pregnancy Childbirth. 2022 Oct 12;22(1):766. doi: 10.1186/s12884-022-05089-w. PMID 36224523